CLINICAL TRIAL: NCT00700297
Title: A Double Blind Cross Over Clinical Trial to Determine Colchicine Efficacy in Behcet's Disease
Brief Title: Colchicine Randomized Double-Blind Controlled Crossover Study in Behcet's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Fereydoun Davatchi, Head Rheumatology Research Center, Rheumatology Research Center, Tehran University for Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rrc-23
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-05

CONDITIONS: Behcet's Syndrome
Keywords: Oral aphthosis; Genital aphthosis; Psuedofolliculitis; Erythem nodusom; Joint manifestations; Colchicine
MeSH Terms: conditions — Behcet Syndrome | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Active Comparator): Patients who received Colchicine and went on placebo after 4 months
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Patients who received placebo and went on Colchicine after 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — 100 mg Colchicine per day for 4 months
  Other Names: Modacine
  Arms: Colchicine
Drug: Placebo — One tablet placebo per day for 4 months
  Arms: Placebo

SUMMARY:
Colchicine was first used in Behcet's Disease (BD), in 1977. There are controversial reports of the efficacy of Colchicine in BD. For some experts the unresponsiveness of some patients could be explained by genetic difference between the Silk Road BD and sporadic BD from other parts of the world.

To test this hypothesis (the inefficacy of colchicine in the Silk Road BD), we designed a randomized double-blind controlled crossover study in Iran, which is in the middle of the Silk Road, and has the second highest prevalence of BD in the world.

DETAILED DESCRIPTION:
Patients: They were selected as consecutive patients.

The entry criteria was: age between 14 and 60 years, confirmed diagnosis of Behcet's Disease, absence of major organ involvement (eye, brain, lung, and cardio-vascular involvement), having at least one active symptom, and no treatment for at least one month. Patients were explained the study design and they gave a signed written consent. During the two phases of study, if a major organ involvement appeared, the patient was moved out of the study. All patients fulfilled the new International Criteria for Behcet's Disease.

Method: patients were randomized at the study entry to take either colchicine or placebo. At 4 months, they were crossed over. Those who were taking colchicine went on placebo and those on placebo went on colchicine. Each patient tried therefore, both colchicine and placebo. The primary outcome was the effect of colchicine on the disease activity index, the IBDDAM (16-17). To calculate the overall IBDDAM of the baseline, the IBDDAM of the last 12 months (prior to the study) of each manifestation was calculated and added together. The overall disease activity index was then divided to the number of months (12 months) to have the mean activity index per month. IBDDAM was then measured every 2 months (in the middle and at the end, in each arm of the study). The total IBBDAM of the 4 months was then divided by 4 to have the mean activity index per month. The secondary outcome was to see how the individual symptoms responded to colchicine (IBDDAM of each manifestation).

Statistical analysis: The analysis was done by the intention to treat method. As the difference between IBDDAM before and after treatment had normal distribution Student T test for paired samples were used to evaluate the outcome in the colchicine and the placebo group. As the Levene's test showed the homogeneity of variance, ANOVA (one way) was used to test the effect of treatment (colchicine and placebo) and gender on patients' outcome. The dependent variable was the difference between IBDDAM (before and after the treatment). The independent variables were the treatment, and the gender. SPSS 15 was used for all statistical calculations.

ELIGIBILITY:
Inclusion Criteria:

* Patient's who fulfilled the International Criteria for Behcet's Disease.

Exclusion Criteria:

* major organ involvement
* Hypersensitivity reaction

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 169 (Actual)
Dates: Start 2002-08; Primary Completion 2005-10 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Iranian Behcet's Disease Dynamic Activity Measurement (IBDDAM) | 8 months

SECONDARY OUTCOMES:
Oral Aphthosis | 8 months
Genital Aphthosis | 8 months
Psuedofolliculitis | 8 months
Erythem Nodusom | 8 months
Joint Manifestations | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Fereydoun Davatchi, Professor, Study Chair — Rheumatology Research Center, Tehran University for Medical Sciences; Bahar Sadeghi, MD, Principal Investigator — Rheumatology research Center, Tehran University for Medical Sciences; Arash Tehrani Banihashemi, MD, MPH, Principal Investigator — Rheumatology Research Center, Tehran University for Mrdical Sciences; Farhad Shahram, Professor, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences
Locations (1):
- Rheumatology research Center, Tehran UMS, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Davatchi F, Shams H, Rezaipoor M, Sadeghi-Abdollahi B, Shahram F, Nadji A, Chams-Davatchi C, Akhlaghi M, Faezi T, Naderi N. Rituximab in intractable ocular lesions of Behcet's disease; randomized single-blind control study (pilot study). Int J Rheum Dis. 2010 Aug;13(3):246-52. doi: 10.1111/j.1756-185X.2010.01546.x. PMID 20704622
- [Derived] Davatchi F, Sadeghi Abdollahi B, Tehrani Banihashemi A, Shahram F, Nadji A, Shams H, Chams-Davatchi C. Colchicine versus placebo in Behcet's disease: randomized, double-blind, controlled crossover trial. Mod Rheumatol. 2009;19(5):542-9. doi: 10.1007/s10165-009-0200-2. Epub 2009 Jul 14. PMID 19597921